CLINICAL TRIAL: NCT00044031
Title: Prospective, Randomized, Controlled, Double-Blind, Multi-National, Multi-Center Study of G17DT Immunogen in Combination With Gemcitabine Versus Placebo in Combination With Gemcitabine in Previously Untreated Subjects With Locally Advanced (Nonresectable Stage II and III), Recurrent Disease Following Primary Resection, or Metastatic (Stage IV) Adenocarcinoma of the Pancreas (Protocol No. PC4)
Brief Title: Safety and Efficacy of G17DT Immunogen Combined With Gemcitabine vs. Gemcitabine in the Treatment of Advanced Pancreatic Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC4
Expanded Access: Available
Record Dates: First submitted 2002-08-16; First posted 2002-08-20 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; G17DT; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — gastrin immunogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Placebo Comparator): Placebo (immunogen vehicle) combined with gemcitabine.
- A (Experimental): 500 µg G17DT immunogen combined with gemcitabine.
  Interventions: Biological: G17DT Immunogen

INTERVENTIONS:
Biological: G17DT Immunogen
  Arms: A

SUMMARY:
This study will test whether the G17DT Immunogen, when administered in combination with chemotherapy, is an effective and safe treatment for pancreatic cancer.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of pancreatic adenocarcinoma and unsuitable for pancreatic tumor resection
* Life expectancy of at least 3 months
* Functional status by Karnofsky Index of at least 70

Exclusion criteria:

* Prior treatment with chemotherapy, radiotherapy, or anti-cancer immunotherapy
* Chronic use of corticosteroids, except for inhaled corticosteroids used for asthma or chronic obstructive pulmonary disease
* Immunodeficiency
* Bone marrow transplant within past year
* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2001-02; Primary Completion 2004-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Survival | Up to 12 months

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 12 months
  Adverse events, defined as any event involving adverse reactions, illnesses with onset during the study, or exacerbations of pre-existing illnesses, were assessed at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: R Hawkins, M.D., Principal Investigator — Christie Hospital, Manchester